CLINICAL TRIAL: NCT04977687
Title: Using Machine Learning to Predict Acute Kidney Injury Requiring Renal Replacement Therapy After Cardiac Surgery
Brief Title: Machine Learning Predict Renal Replacement Therapy After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yunlong Fan, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: chinaPLAGH-08983219
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Machine Learning; Acute Kidney Injury; Renal Replacement Therapy; Prediction Models
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is a major complication which may result in adverse impact on short- and long-term mortality. The researcher here developed several prediction models based on machine learning technique to allow early identification of patients who at the high risk of unfavorable kidney outcomes. The retrospective study comprised 2108 consecutive patients who underwent cardiac surgery from January 2017 to December 2020.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years who underwent cardiac surgery

Exclusion Criteria:

* data miss greater than 10%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age over 18 years who underwent cardiac surgery
Sampling Method: Probability Sample
Enrollment: 2108 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
patients required renal replacement therapy | 14 days
  The primary outcome was patients with the requirement for acute dialysis within 14 days after cardiac surgery. Renal replacement therapy is recommended for patients with severe acute kidney injury as well as hemodynamic instability or severe electrolyte disturbances (e.g. blood potassium > 6) or acid-base balance disturbances (e.g. H value less than or equal to 7.15).
  Prior to the start of renal replacement therapy, the investigator invited a consultation with the nephrology department to assess the condition

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General hospital, Beijing, Beijing Municipality, China